CLINICAL TRIAL: NCT03024281
Title: Surveillance of Azole Resistance in Aspergillus
Brief Title: Surveillance of Azole Resistance in Aspergillus Isolates in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 201605098RIPA
Record Dates: First submitted 2016-11-21; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Infection; Aspergillus
Keywords: Aspergillus; Antifungal susceptibility; Azole resistance
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary objectives:

1. To investigate the prevalence of azole resistance in Aspergillus clinical isolates collected in participating hospitals in Taiwan
2. To investigate the prevalence of azole resistance in Aspergillus environmental isolates in Taiwan
3. To characterize the molecular mechanisms of azole resistance in Aspergillus isolates in Taiwan
4. To investigate the clonality of Aspergillus clinical and environmental isolates in Taiwan
5. To describe the genetic relationships between local resistant strains with global strains

Secondary objective:

1. To describe the clinical characteristics and treatment outcome of patients with proven or probable invasive aspergillosis
2. To evaluate the clinical impact of azole resistance in patients with proven or probable invasive aspergillosis in a case-control study

DETAILED DESCRIPTION:
Cumulative evidence described the emergence and geographical expansion of azole-resistant Aspergillus fumigatus associated with azole treatment failure. Multiple amino acid substitutions in the cyp51A gene have been described to be associated with azole resistance that emerges during azole treatment, while a resistance mechanism, TR34/L98H mutation in cyp51A, has been linked to the agricultural use of azole fungicides in Europe, which have also been widely used in Taiwan for years. The current prevalence of azole-resistant Aspergillus isolates and mechanisms of azole resistance in Taiwan is not clear. Considering the potential of geographic migration of resistant isolates from neighboring countries and the possibility of emergence of locally revolved resistant strains, this 2-year multi-center project aims to investigate the prevalence rate of azole resistance in Aspergillus clinical and environmental isolates, to determine the molecular mechanisms of azole resistance, and to describe the clinical characteristics and treatment outcome of Aspergillus diseases in Taiwan. Clinical and environmental Aspergillus isolates will be collected and examined, and clinical data from patients with Aspergillus diseases or colonization will be retrieved and analyzed. Through this study the investigators anticipate increase in awareness of prevalence and impact of azole resistance in patient safety in participating hospitals. In addition, the investigators may update Taiwan treatment guideline for aspergillosis on the basis of these evidence and knowledge.

ELIGIBILITY:
For primary objectives

Inclusion Criteria:

* Patients with one or more clinical specimens culture positive of Aspergillus

Exclusion Criteria:

* Is not a human pathogen of Aspergillus
* no clinical data available

For secondary objectives (a case-control study in a 1:4 ratio)

Inclusion Criteria:

* patients with proven or probable invasive aspergillosis

Case patients: patients infected by azole-resistant isolates Control patients: patients infected by azole-susceptible isolates

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 10 hospitals located in different geographic location of Taiwan will be invited to participate this project. These hospitals are selected based on three criteria: better quality of routine microbiology laboratory (not reference laboratory), one or more physicians or microbiologists who are interested in medical mycology, and geographic location of the hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 6 weeks after diagnosis of proven or probable invasive aspergillosis
  The proportion of patients with complete response or partial response according to the definition described in "Segal BH, Herbrecht R, Stevens DA, Ostrosky-Zeichner L, Sobel J, Viscoli C, et al. Defining responses to therapy and study outcomes in clinical trials of invasive fungal diseases: Mycoses Study Group and European Organization for Research and Treatment of Cancer consensus criteria. Clin Infect Dis. Sep 1 2008;47(5):674-683."

SECONDARY OUTCOMES:
All-cause mortality | 6 weeks after diagnosis of proven or probable invasive aspergillosis
  The proportion of non-survivors. Discharge against medical advice and in critical condition and lost to follow up will categorized as mortality.
All-cause mortality | 12 weeks after diagnosis of proven or probable invasive aspergillosis
  The proportion of non-survivors. Discharge against medical advice and in critical condition and lost to follow up will categorized as mortality.
Breakthrough mold infections | 6 weeks after diagnosis of proven or probable invasive aspergillosis
  The proportion of patients with breakthrough mold infections
Breakthrough invasive fungal diseases | 12 weeks after diagnosis of proven or probable invasive aspergillosis
  The proportion of patients with breakthrough invasive fungal diseases defined as occurrence of a proven or probable invasive fungal diseases according to EORTC/MSG revised definitions while on systemic antifungal therapy or within 15 days of discontinuation of antifungal use
Treatment success | 12 weeks after diagnosis of proven or probable invasive aspergillosis
  The proportion of patients with complete response or partial response.

CONTACTS AND LOCATIONS:
Overall Officials: WHO, ICMJE WHO and ICMJE, Study Director — WHO and ICMJE
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided